CLINICAL TRIAL: NCT01667133
Title: A Phase 1/2 Multi-center, Open-label Study of Ponatinib in Japanese Patients With Chronic Myeloid Leukemia (CML) Who Have Failed Dasatinib or Nilotinib or Ph+ Acute Lymphoblastic Leukemia (ALL) Who Have Failed Prior Tyrosine Kinase Inhibitors (TKIs)
Brief Title: A Study of Ponatinib in Japanese Participants With Chronic Myeloid Leukemia (CML) and Ph+ Acute Lymphoblastic Leukemia (ALL)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ariad Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AP24534-11-106
Record Dates: First submitted 2012-08-13; First posted 2012-08-17 (Estimated); Results first posted 2022-06-13 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-03

CONDITIONS: Chronic Myeloid Leukemia (CML); Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia (Ph+ ALL)
Keywords: Leukemia; Leukemia, Myeloid; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Neoplasms by Histologic Type; Neoplasms; Lymphoproliferative Disorders; Lymphatic Diseases; Immunoproliferative Disorders; Immune System Diseases; Myeloproliferative Disorders; Bone Marrow Diseases; Hematologic Diseases
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia; Leukemia, Myeloid; Neoplasms by Histologic Type; Neoplasms; Lymphoproliferative Disorders; Lymphatic Diseases; Immunoproliferative Disorders; Immune System Diseases; Myeloproliferative Disorders; Bone Marrow Diseases; Hematologic Diseases | interventions — ponatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phase 1 dose escalation (Experimental): Phase 1
  Interventions: Drug: ponatinib - Phase 1
- Phase 2 expansion (Experimental): Phase 2
  Interventions: Drug: ponatinib - Phase 2

INTERVENTIONS:
Drug: ponatinib - Phase 1 — 30 mg dose of ponatinib taken orally once daily for at least the first 6 patients. If no dose-limiting toxicities are observed, the next patients will receive 45 mg dose of ponatinib taken orally once daily. Once the recommended dose is confirmed, all patients may receive the recommended dose, at the investigators' discretion.
  Other Names: AP24534
  Arms: Phase 1 dose escalation
Drug: ponatinib - Phase 2 — Recommended dose of ponatinib as determined in the dose escalation phase. In addition, 3 patients will receive 15 mg dose once daily for 8 days for PK testing. These PK patients may be allowed to receive the recommended dose after PK testing is complete, at the investigators' discretion.
  Other Names: AP24534
  Arms: Phase 2 expansion

SUMMARY:
The purpose of this study is to assess the safety and efficacy of ponatinib in Japanese patients with chronic myeloid leukemia (CML) who have experienced failure of dasatinib or nilotinib or with Ph+ acute lymphoblastic leukemia (ALL) following failure of prior tyrosine kinase inhibitors (TKIs).

DETAILED DESCRIPTION:
This multi-center, phase 1/2, open-label study will consist of two phases. The first will be a dose escalation phase employing a modified 3+3 design with two dose cohorts (30mg and 45mg). After 6 patients complete the first cycle in a cohort, safety events will be evaluated before opening the next dose cohort. Patients will continue on treatment as long as it is tolerated and disease progression has not occurred. Phase 2 will occur at the recommended dose determined in phase 1 in an additional 25 patients. Another 3 patients will be dosed at 15mg for collection of pharmacokinetic data. These patients may also escalate to the recommended dose and be assessed for efficacy and safety as phase 2 patients.

Efficacy measures include molecular, cytogenetic, and hematologic response rates at various time points; time to response; duration of response; and survival follow-up. Safety measures include routine physical and laboratory evaluations, adverse event monitoring, and ECGs. Other measures include mutation testing and molecular genetic assessment. Accrual is expected to take approximately 12 months, and patients will be followed for survival for up to 60 months from the last dose of study drug; therefore, the estimated duration of the trial is 72 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have CML in any phase (CP, AP, or BP of any phenotype) or Ph+ ALL, as follows:

   * All patients must have screening bone marrow (BM) cytogenetics with conventional banding performed within 42 days prior to beginning treatment.
   * Examination of at least 20 metaphases is required in patients in CP. If less than 20 metaphases are examined, the BM aspirate must be repeated.
   * Adequate BM aspirate with differential cell counts is required in patients with AP, BP, or Ph+ ALL. If an adequate aspirate is not obtained, the aspirate must be repeated.
2. Be previously treated with and resistant, or intolerant, as defined in the protocol, to either dasatinib or nilotinib for CML or at least one TKI for Ph+ ALL, regardless of whether dasatinib or nilotinib or the prior TKI were used to treat newly diagnosed or resistant patients.
3. Must be ≥ 18 years old.
4. Provide written informed consent.
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
6. Minimum life expectancy of 3 months or more.
7. Adequate renal function defined as serum creatinine < 1.5 × upper limit of normal (ULN) for institution.
8. Adequate hepatic function defined as:

   1. Total bilirubin < 1.5 × ULN
   2. Alanine aminotransferase (ALT [SGPT]) and aspartate aminotransferase (AST [SGOT]) < 2.5 × ULN for institution (< 5 × ULN if liver involvement with leukemia)
   3. Prothrombin time < 1.5 × ULN
9. Normal pancreatic status defined as:

   1. Lipase ≤ 1.5 × ULN for institution
   2. Amylase ≤ 1.5 × ULN for institution
10. Normal QT interval corrected (Fridericia) (QTcF) interval on screening ECG evaluation, defined as QTcF of ≤ 450 ms in males or ≤ 470 ms in females.
11. For females of childbearing potential, a negative pregnancy test must be documented prior to enrolment.
12. Female and male patients who are of childbearing potential must agree to use an effective form of contraception with their sexual partners throughout participation in this study.
13. Ability to comply with study procedures, in the Investigator's opinion.

Exclusion Criteria:

Patients are not eligible for participation in the study if they meet any of the following exclusion criteria:

1. Received TKI therapy within 7 days prior to receiving the first dose of ponatinib, or have not recovered (> grade 1 by National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.0 [NCI CTCAE v.4.0]) from adverse events (AEs) (except alopecia) due to agents previously administered.
2. Received other therapies as follows:

   1. For CP and AP patients, received interferon, cytarabine, or immunotherapy within 14 days, or any other cytotoxic chemotherapy, radiotherapy, or investigational therapy within 28 days prior to receiving the first dose of ponatinib.
   2. For BP patients, received chemotherapy within 7 days prior to the first dose of ponatinib. Otherwise, 2a applies.
   3. For Ph+ ALL patients, received corticosteroids within 24 hours before the first dose of ponatinib and other chemotherapy within 7 days prior to the first dose of ponatinib. Otherwise, 2a applies.
   4. All patients are excluded if they have not recovered (> grade 1 by NCI CTCAE v.4.0) from AEs (except alopecia) due to agents previously administered.
3. Underwent autologous or allogeneic stem cell transplant < 60 days prior to receiving the first dose of ponatinib; any evidence of ongoing graft versus-host disease (GVHD) or GVHD requiring immunosuppressive therapy.
4. Take medications that are known to be associated with Torsades de Pointes.
5. Require concurrent treatment with immunosuppressive agents, other than corticosteroids prescribed for a short course of therapy.
6. Have previously been treated with ponatinib.
7. Patients with CP-CML are excluded if they are in CCyR.
8. Patients with CP-CML are excluded if a baseline BM aspirate adequate for conventional cytogenetic analysis with 20 metaphases examined is not available.
9. Patients with AP-CML, BP-CML, or Ph+ ALL are excluded if they are in MaHR.
10. Patients with AP-CML, BP-CML, or Ph+ ALL are excluded if a baseline BM aspirate adequate for cell count and differential report is not available. Patients with a fibrotic marrow or dry tap that does not yield adequate cell counts for diagnosis are not evaluable for classification, and endpoints are not eligible.
11. Have active central nervous system (CNS) disease as evidenced by cytology or pathology. In the absence of clinical CNS disease, lumbar puncture is not required. History itself of CNS involvement is not exclusionary if CNS has been cleared with a documented negative lumbar puncture.
12. Have significant or active cardiovascular disease, specifically including, but not restricted to:

    1. Myocardial infarction within 3 months prior to first dose of ponatinib
    2. History of clinically significant atrial arrhythmia or any ventricular arrhythmia
    3. Unstable angina within 3 months prior to first dose of ponatinib
    4. Congestive heart failure within 3 months prior to first dose of ponatinib
13. Have a significant bleeding disorder unrelated to CML or Ph+ ALL.
14. Have a history of pancreatitis or alcohol abuse.
15. Have uncontrolled hypertriglyceridemia (triglycerides > 450 mg/dL).
16. Have malabsorption syndrome or other gastrointestinal illness that could affect absorption of orally administered ponatinib.
17. Have been diagnosed with another primary malignancy within the past 3 years (except for non-melanoma skin cancer or cervical cancer in situ, or controlled prostate cancer, which are allowed within 3 years).
18. Are pregnant or lactating. Women of childbearing potential must agree to an effective contraception from the time of signing the informed consent through the Follow-up Visit, approximately 30 days after last dose of ponatinib.
19. Underwent major surgery (with the exception of minor surgical procedures, such as catheter placement or BM biopsy) within 14 days prior to first dose of ponatinib.
20. Have ongoing or active infection (including known history of human immunodeficiency virus [HIV], hepatitis B virus [HBV], or hepatitis C virus [HCV]). Testing for these viruses is not required in the absence of history.
21. Suffer from any condition or illness that, in the opinion of the Investigator or the Medical Monitor, would compromise patients safety or interfere with the evaluation of the safety of the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-08-31 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2018-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (11):
- Japan (11):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - Akita University Hospital, Akita, Akita
  - Hiroshima Red Cross Hospital & Atomic-bomb Survivors Hospital, Hiroshima, Hiroshima
  - Kyushu University Hospital, Hukuoka-shi, Hukuoka
  - Kinki University Hospital, Faculty of Medicine, Osakasayama-shi, Osaka
  - The Cancer Institute Hospital Japanese Foundation for Cancer Research, Koto, Tokyo
  - The University of Tokyo, The Institute of Medical Science, Minato-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Osaka City University Hospital, Shinjuku-ku, Tokyo
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Tokyo Medical University Hospital, Shinjuku-ku, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Hanley MJ, Diderichsen PM, Narasimhan N, Srivastava S, Gupta N, Venkatakrishnan K. Population Pharmacokinetics of Ponatinib in Healthy Adult Volunteers and Patients With Hematologic Malignancies and Model-Informed Dose Selection for Pediatric Development. J Clin Pharmacol. 2022 Apr;62(4):555-567. doi: 10.1002/jcph.1990. Epub 2021 Dec 16. PMID 34699069
- [Derived] Tojo A, Kyo T, Yamamoto K, Nakamae H, Takahashi N, Kobayashi Y, Tauchi T, Okamoto S, Miyamura K, Hatake K, Iwasaki H, Matsumura I, Usui N, Naoe T, Tugnait M, Narasimhan NI, Lustgarten S, Farin H, Haluska F, Ohyashiki K. Ponatinib in Japanese patients with Philadelphia chromosome-positive leukemia, a phase 1/2 study. Int J Hematol. 2017 Sep;106(3):385-397. doi: 10.1007/s12185-017-2238-9. Epub 2017 Apr 25. PMID 28444644

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 9 investigative sites in Japan from 31 August 2012 to 02 August 2018.
Pre-assignment Details: Participants with CP-CML, AP-CML, or BP-CML, or with Ph+ALL were enrolled in Phase 1 (dose-escalation) to receive 30 or 45 mg of ponatinib and recommended phase 2 dose in Phase 2 (expansion). As there was no participant enrolled in Phase 1: BP-CML Ponatinib 30 milligram (mg) arm, therefore the arm is not reported in the result summary. Participants in Phase 1 with CP-CML or AP-CML, BP-CML or Ph+ ALL and who had T315I mutation and other mutations were analyzed as subgroups in the study.
Groups:
- Ponatinib 30 mg: Phase 1 CP-CML: Ponatinib 30 mg, tablet, orally, once daily in a 28-day treatment cycle for up to unacceptable drug reaction or disease progression (up to 60 months) in participants with chronic phase (CP)-chronic myeloid leukemia (CML) resistant or intolerant to dasatinib or nilotinib in Dose-escalation Phase 1.
- Ponatinib 30 mg: Phase 1 AP-CML: Ponatinib 30 mg, tablet, orally, once daily in a 28-day treatment cycle for up to unacceptable drug reaction or disease progression (up to 60 months) in participants with accelerated phase (AP)- CML resistant or intolerant to dasatinib or nilotinib in Dose-escalation Phase 1.
- Ponatinib 30 mg: Phase 1 Ph+ ALL: Ponatinib 30 mg, tablet, orally, once daily in a 28-day treatment cycle for up to unacceptable drug reaction or disease progression (up to 60 months) in participants with Philadelphia chromosome plus acute lymphoblastic leukemia (Ph+ ALL) resistant or intolerant to prior tyrosine kinase inhibitor (TKIs) in Dose-escalation Phase 1.
- Ponatinib 45 mg: Phase 1 CP-CML: Ponatinib 45 mg, tablet, orally, once daily in a 28-day treatment cycle for up to unacceptable drug reaction or disease progression (up to 60 months) in participants with CP-CML resistant or intolerant to dasatinib or nilotinib in Dose-escalation Phase 1.
- Ponatinib 45 mg: Phase 1 AP-CML: Ponatinib 45 mg, tablet, orally, once daily in a 28-day treatment cycle 1 for up to unacceptable drug reaction or disease progression (up to 60 months) in participants with AP-CML resistant or intolerant to dasatinib or nilotinib in Dose-escalation Phase 1.
- Ponatinib 45 mg: Phase 1 BP-CML: Ponatinib 45 mg, tablet, orally, once daily in a 28-day treatment cycle for up to unacceptable drug reaction or disease progression (up to 60 months) in participants with BP-CML resistant or intolerant to dasatinib or nilotinib in Dose-escalation Phase 1.
- Ponatinib 45 mg: Phase 1 Ph+ ALL: Ponatinib 45 mg, tablet, orally, once daily in a 28-day treatment cycle for up to unacceptable drug reaction or disease progression (up to 60 months) in participants with Ph+ ALL resistant or intolerant to prior TKIs in Dose-escalation Phase 1.
- Ponatinib 15 mg: Phase 2 CP- CML: Ponatinib 15 mg, tablet, orally, once daily for 7-days in a 28-day treatment cycle in participants with CP-CML resistant or intolerant to dasatinib or nilotinib in Expansion Phase 2. Dose was increased to ponatinib 45 mg in the same participants at the discretion of Investigator and was administered as tablet, orally, once daily in a 28-day treatment cycle for up to unacceptable drug reaction or disease progression (up to 60 months).
- Ponatinib 15 mg: Phase 2 Ph+ ALL: Ponatinib 15 mg, tablet, orally, once daily for 7-days in a 28-day treatment cycle in participants with Ph+ ALL resistant or intolerant to prior TKIs in Expansion Phase 2. Dose was increased to ponatinib 45 mg in the same participants at the discretion of Investigator and was administered as tablet, orally, once daily in a 28-day treatment cycle 1 for up to unacceptable drug reaction or disease progression (up to 60 months).
- Ponatinib 45 mg: Phase 2 CP-CML: Ponatinib 45 mg, tablet, orally, once daily in a 28-day treatment cycle for up to unacceptable drug reaction or disease progression (up to 60 months) in participants with CP-CML resistant or intolerant to dasatinib or nilotinib in Expansion Phase 2.
- Ponatinib 45 mg: Phase 2 BP-CML: Ponatinib 45 mg, tablet, orally, once daily in a 28-day treatment cycle for up to unacceptable drug reaction or disease progression (up to 60 months) in participants with BP-CML resistant or intolerant to dasatinib or nilotinib in Expansion Phase 2.
- Ponatinib 45 mg: Phase 2 PH+ ALL: Ponatinib 45 mg, tablet, orally, once daily in a 28-day treatment cycle for up to unacceptable drug reaction or disease progression (up to 60 months) in participants with PH+ ALL resistant or intolerant to prior TKI in Expansion Phase 2.
Period: Phase 1: Dose-escalation
Arm/Group | Ponatinib 30 mg: Phase 1 CP-CML | Ponatinib 30 mg: Phase 1 AP-CML | Ponatinib 30 mg: Phase 1 Ph+ ALL | Ponatinib 45 mg: Phase 1 CP-CML | Ponatinib 45 mg: Phase 1 AP-CML | Ponatinib 45 mg: Phase 1 BP-CML | Ponatinib 45 mg: Phase 1 Ph+ ALL | Ponatinib 15 mg: Phase 2 CP- CML | Ponatinib 15 mg: Phase 2 Ph+ ALL | Ponatinib 45 mg: Phase 2 CP-CML | Ponatinib 45 mg: Phase 2 BP-CML | Ponatinib 45 mg: Phase 2 PH+ ALL
Started | 1 | 1 | 4 | 3 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Completed | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 4 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 0 | 1 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 2: Dose-expansion
Arm/Group | Ponatinib 30 mg: Phase 1 CP-CML | Ponatinib 30 mg: Phase 1 AP-CML | Ponatinib 30 mg: Phase 1 Ph+ ALL | Ponatinib 45 mg: Phase 1 CP-CML | Ponatinib 45 mg: Phase 1 AP-CML | Ponatinib 45 mg: Phase 1 BP-CML | Ponatinib 45 mg: Phase 1 Ph+ ALL | Ponatinib 15 mg: Phase 2 CP- CML | Ponatinib 15 mg: Phase 2 Ph+ ALL | Ponatinib 45 mg: Phase 2 CP-CML | Ponatinib 45 mg: Phase 2 BP-CML | Ponatinib 45 mg: Phase 2 PH+ ALL
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 11 | 3 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 6 | 3 | 6
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated population included all participants who had received at least 1 dose of study drug.
Groups:
- Ponatinib 30 mg: Phase 1 CP-CML: Ponatinib 30 mg, tablet, orally, once daily in a 28-day treatment cycle for up to unacceptable drug reaction or disease progression (up to 60 months) in participants with CP-CML resistant or intolerant to dasatinib or nilotinib in Dose-escalation Phase 1.
- Ponatinib 30 mg: Phase 1 AP-CML: Ponatinib 30 mg, tablet, orally, once daily in a 28-day treatment cycle for up to unacceptable drug reaction or disease progression (up to 60 months) in participants with AP-CML resistant or intolerant to dasatinib or nilotinib in Dose-escalation Phase 1.
- Ponatinib 30 mg: Phase 1 Ph+ ALL: Ponatinib 30 mg, tablet, orally, once daily in a 28-day treatment cycle for up to unacceptable drug reaction or disease progression (up to 60 months) in participants with Ph+ ALL resistant or intolerant to prior TKIs in Dose-escalation Phase 1.
- Ponatinib 15 mg: Phase 2 CP-CML: Ponatinib 15 mg, tablet, orally, once daily for 7-days in a 28-day treatment cycle in participants with CP-CML resistant or intolerant to dasatinib or nilotinib in Expansion Phase 2. Dose was increased to ponatinib 45 mg in the same participants at the discretion of Investigator and was administered as tablet, orally, once daily in a 28-day treatment Cycle for up to unacceptable drug reaction or disease progression (up to 60 months).
- Total: Total of all reporting groups
Arm/Group | Ponatinib 30 mg: Phase 1 CP-CML | Ponatinib 30 mg: Phase 1 AP-CML | Ponatinib 30 mg: Phase 1 Ph+ ALL | Ponatinib 45 mg: Phase 1 CP-CML | Ponatinib 45 mg: Phase 1 AP-CML | Ponatinib 45 mg: Phase 1 BP-CML | Ponatinib 45 mg: Phase 1 Ph+ ALL | Ponatinib 15 mg: Phase 2 CP-CML | Ponatinib 15 mg: Phase 2 Ph+ ALL | Ponatinib 45 mg: Phase 2 CP-CML | Ponatinib 45 mg: Phase 2 BP-CML | Ponatinib 45 mg: Phase 2 PH+ ALL | Total
Number analyzed (Participants) | 1 | 1 | 4 | 3 | 1 | 1 | 1 | 2 | 1 | 11 | 3 | 6 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 | 62.0 | 56.5 (11.73) | 60.7 (12.86) | 57.0 | 58.0 | 30.0 | 61.5 (14.85) | 76.0 | 59.1 (13.78) | 67.7 (4.04) | 58.3 (13.78) | 59.4 (12.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 6 | 1 | 4 | 15
  Male | 1 | 0 | 2 | 3 | 1 | 0 | 1 | 2 | 1 | 5 | 2 | 2 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 1 | 4 | 3 | 1 | 1 | 1 | 2 | 1 | 11 | 3 | 6 | 35
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 1 | 1 | 4 | 3 | 1 | 1 | 1 | 2 | 1 | 11 | 3 | 6 | 35
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 67.0 | 57.0 | 45.8 (3.93) | 74.1 (6.49) | 55.8 | 60.0 | 54.6 | 60.0 (8.49) | 60.5 | 59.0 (9.93) | 54.0 (10.99) | 53.7 (11.84) | 57.5 (10.54)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 163.6 | 155.9 | 165.1 (8.89) | 172.4 (6.61) | 170.5 | 156.4 | 170.7 | 169.5 (2.83) | 166.0 | 159.5 (10.15) | 162.4 (6.92) | 158.0 (8.95) | 162.5 (8.95)
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG performance status used by doctors/researchers to assess how participant's disease is progressing, assess how disease affects daily living activities of participant and determine appropriate treatment/prognosis on 5-point scale. 0=Actively able to do activities; 1=Restricted in physical activity, able to do light/sedentary work; 2=Ambulatory (>50% of waking hours), capable of self-care, unable to do any work activities; 3=Capable of limited self-care, confined to bed >50% of waking hours; 4=Completely disabled, cannot do any self-care, totally confined to bed; 5=dead.
  Participants
    0 = Fully Active | 1 | 1 | 2 | 3 | 0 | 1 | 0 | 2 | 0 | 11 | 1 | 6 | 28
    1 = Restricted in Physical Activity; Ambulatory | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 7
Participants with Initial Diagnosis of Leukemia [Count of Participants; unit: Participants]
  CP-CML | 1 | 1 | 0 | 3 | 1 | 0 | 0 | 2 | 0 | 11 | 1 | 0 | 20
  AP-CML | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  BP-CML | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Ph+ ALL | 0 | 0 | 4 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 6 | 12
Time Since Diagnosis to Date of First Dose [Median (Full Range); unit: years] | 10.29 [10.29 to 10.29] | 21.65 [21.65 to 21.65] | 1.51 [1.28 to 9.64] | 3.47 [0.46 to 20.04] | 10.87 [10.87 to 10.87] | 0.53 [0.53 to 0.53] | 3.00 [3.00 to 3.00] | 12.98 [0.36 to 25.60] | 0.73 [0.73 to 0.73] | 3.76 [0.96 to 17.11] | 1.69 [0.25 to 6.05] | 0.91 [0.24 to 2.11] | 2.11 [0.24 to 25.60]
Participants with Extramedullary Involvement [Count of Participants; unit: Participants] — Participants with extramedullary disease sites were assessed. Extramedullary disease occurs when myeloma cells form tumors outside the bone marrow in the soft tissues or organs of the body.
  Participants
    Hepatomegaly | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
    Splenomegaly | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    No extramedullary involvement | 1 | 1 | 4 | 3 | 0 | 1 | 1 | 2 | 1 | 11 | 2 | 6 | 33
Participants with BCR-ABL Ratio [Count of Participants; unit: Participants] — Breakpoint cluster region-Abelson complex (BCR-ABL1) is an abnormal gene found in CML and acute lymphoblastic leukemia (ALL). The chromosomal defect in the Philadelphia chromosome is a translocation, in which parts of two chromosomes, 9 and 22, swap places. The result is that a fusion gene is created by juxtapositioning the Abl1 gene on chromosome 9 to a part of the BCR gene on chromosome 22. Depending upon the breakpoints on the BCR gene, there are several forms of fusion proteins. BCR-ABL ratio is assessed in % international scale (IS).
  Participants
    Greater than (>)0.1 - less than or equal to (<=)1% | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 3
    >1 to <=10 percent (%) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 3
    >10% | 1 | 1 | 1 | 2 | 1 | 1 | 0 | 1 | 0 | 7 | 2 | 2 | 19
    e1a2 variant | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants With Dose-limiting Toxicities (DLTs) as a Measure of Safety Profile to Determine Recommended Dose of Ponatinib
Description: DLT was evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0 and was defined as any of the following events: 1. Grade greater than or equal to (>=) 3 non-hematologic, with the exception of medically controllable toxicities (example; nausea, vomiting, fatigue, electrolyte disturbances, hypersensitivity reactions) lasting <=3 days, but excluding alopecia; 2. Missed doses: >25% of planned ponatinib doses over 28 days due to AEs in the first cycle; 3. Febrile neutropenia (the occurrence of an ANC <500/microliter concurrently with a temperature elevation of >101 degree Fahrenheit), when neutropenia is not related to underlying acute leukemia, as defined hematologic toxicity: Dose-limiting hematologic toxicity is the occurrence of a Grade 4 cytopenia >28 days, not related to underlying disease according to the investigator. Bone marrow examination must demonstrate <5% cellularity.
Time Frame: Cycle 1 (Cycle length= 28 days)
Population: DLT evaluable population (Phase 1 only) included all participants who had completed at least 75% of their planned doses during Cycle 1, unless missed doses were due to adverse events (AEs).
Measure: Count of Participants; unit: Participants
Groups:
- Ponatinib 45 mg: Phase 1 AP CML: Ponatinib 45 mg, tablet, orally, once daily in a 28-day treatment cycle 1 for up to unacceptable drug reaction or disease progression (up to 60 months) in participants with AP-CML resistant or intolerant to dasatinib or nilotinib in Dose-escalation Phase 1.
Arm/Group | Ponatinib 30 mg: Phase 1 CP-CML | Ponatinib 30 mg: Phase 1 AP-CML | Ponatinib 30 mg: Phase 1 Ph+ ALL | Ponatinib 45 mg: Phase 1 CP-CML | Ponatinib 45 mg: Phase 1 AP CML | Ponatinib 45 mg: Phase 1 BP-CML | Ponatinib 45 mg: Phase 1 Ph+ ALL
Number analyzed (Participants) | 1 | 1 | 4 | 3 | 1 | 1 | 1
Participants | 0 | 0 | 1 | 1 | 0 | 0 | 0

2. Primary Outcome: Phase 2, CP-CML Participants: Percentage of Participants With Major Cytogenetic Response (MCyR)
Description: MCyR was defined as percentage of participants who achieved a complete cytogenetic response (CCyR) or partial cytogenetic response (PCyR) after the initiation of study treatment. Cytogenic response was the percentage of Philadelphia chromosome positive (Ph+) metaphases in bone marrow. CCyR: no Ph+ cells. PCyR: 1% to 35% Ph+ cells. Participants entering the study already in PCyR had to achieve a CCyR in order to be considered a success for the confirmed MCyR rate.
Time Frame: Baseline up to 60 months
Population: Treated population included all participants who had received at least 1 dose of study drug. This outcome measure was planned to be assessed only in CP-CML participants of Phase 2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ponatinib 15 mg: Phase 2 CP-CML | Ponatinib 45 mg: Phase 2 CP-CML
Number analyzed (Participants) | 2 | 11
percentage of participants | 50 [1.3 to 98.7] | 63.6 [30.8 to 89.1]

3. Primary Outcome: Phase 2, BP-CML and Ph+ALL: Percentage of Participants With Major Hematologic Response (MaHR)
Description: MaHR was defined as percentage of participants with complete hematologic response (CHR) or no evidence of leukemia (NEL). MaHR response was confirmed by a peripheral blood complete blood count (CBC) and differential no earlier than 28 days after the response was observed. Response criteria for CHR was reported as white blood cells (WBC)<=institutional upper limit of normal (ULN), absolute neutrophil count (ANC)>=1000/mm^3, platelets>=100,000/mm^3, no blasts or promyelocytes in peripheral blood, BM blasts <=5%, <5% myelocytes plus metamyelocytes in peripheral blood, basophils in peripheral blood <5%, no extramedullary involvement; Response criteria for NEL reported as WBC<=institutional ULN, no blasts or promyelocytes in peripheral blood, BM blasts <=5%, <5% myelocytes plus metamyelocytes in peripheral blood, basophils in peripheral blood <5%, no extramedullary involvement, at least 1 of the following: (i) 20,000/mm^3<=platelets<100,000/mm^3; (ii) 500/mm^3<=ANC<1000/mm^3.
Time Frame: Baseline up to 60 months
Population: Treated population included all participants who had received at least 1 dose of study drug. This outcome measure was planned to be assessed only in BP-CML and Ph+ALL participants of Phase 2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ponatinib 15 mg: Phase 2 Ph+ ALL | Ponatinib 45 mg: Phase 2 BP-CML | Ponatinib 45 mg: Phase 2 PH+ ALL
Number analyzed (Participants) | 1 | 3 | 6
percentage of participants | 0 [0 to 97.5] | 33.3 [0.8 to 90.6] | 83.3 [35.9 to 99.6]

4. Secondary Outcome: CP-CML Participants: Percentage of Participants With CHR
Description: Hematologic response was defined as CHR for CP-CML participants. Participants who entered the trial in CHR and continued to meet the criteria for CHR on study were analyzed as responders. Response criteria for CHR was reported as WBC <=institutional ULN, platelets <450,000 per cubic millimeter (/mm^3), no blasts or promyelocytes in peripheral blood, <5% myelocytes plus metamyelocytes in peripheral blood, basophils in peripheral blood <5%, no extramedullary involvement (including no hepatomegaly or splenomegaly).
Time Frame: Baseline up to 60 months
Population: Treated population included all participants who had received at least 1 dose of study drug. This outcome measure was planned to be assessed only in CP-CML Participants of Phase 1 and 2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ponatinib 30 mg: Phase 1 CP-CML | Ponatinib 45 mg: Phase 1 CP-CML | Ponatinib 15 mg: Phase 2 CP-CML | Ponatinib 45 mg: Phase 2 CP-CML
Number analyzed (Participants) | 1 | 3 | 2 | 11
percentage of participants | 100 [2.5 to 100] | 100 [29.2 to 100] | 100 [15.8 to 100] | 90.9 [58.7 to 99.8]

5. Secondary Outcome: CP-CML, AP-CML, BP-CML, and Ph+ALL Participants: Percentage of Participants With Confirmed MCyR
Description: Confirmed MCyR was defined as 2 assessments of CCyR or PCyR at least 28 days apart. Participants entering the trial in PCyR must achieve two consecutive assessments of CCyR no fewer than 28 days apart in order to be considered as meeting the criteria for confirmed MCyR. Participants entering the trial in less than PCyR must achieve two consecutive assessments of PCyR or CCyR no fewer than 28 days apart in order to be considered as meeting the criteria for confirmed MCyR. CCyR: no Ph+ cells. PCyR: 1% to 35% Ph+ cells.
Time Frame: Baseline up to 60 months
Population: Treated population included all participants who had received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Ponatinib 45 mg: Phase 1 Ph+ ALL: Ponatinib 45 mg, tablet, orally, once daily in a 28-day treatment cycle 1 in participant with Ph+ ALL resistant or intolerant to prior TKIs in Dose-escalation Phase 1.
- Ponatinib 45 mg: Phase 2 BP-CML: Ponatinib 45 mg, tablet, orally, once daily in a 28-day treatment cycle for up to unacceptable drug reaction or disease progression (up to 6 months) in participants with BP-CML resistant or intolerant to dasatinib or nilotinib in Expansion Phase 2.
Arm/Group | Ponatinib 30 mg: Phase 1 CP-CML | Ponatinib 30 mg: Phase 1 AP-CML | Ponatinib 30 mg: Phase 1 Ph+ ALL | Ponatinib 45 mg: Phase 1 CP-CML | Ponatinib 45 mg: Phase 1 AP-CML | Ponatinib 45 mg: Phase 1 BP-CML | Ponatinib 45 mg: Phase 1 Ph+ ALL | Ponatinib 15 mg: Phase 2 CP-CML | Ponatinib 15 mg: Phase 2 Ph+ ALL | Ponatinib 45 mg: Phase 2 CP-CML | Ponatinib 45 mg: Phase 2 BP-CML | Ponatinib 45 mg: Phase 2 PH+ ALL
Number analyzed (Participants) | 1 | 1 | 4 | 3 | 1 | 1 | 1 | 2 | 1 | 11 | 3 | 6
percentage of participants | 100 [2.5 to 100] | 0 [0.0 to 97.5] | 0 [0 to 60.2] | 100 [29.2 to 100] | 100 [2.5 to 100] | 100 [2.5 to 100] | 100 [2.5 to 100] | 0 [0.0 to 84.2] | 0 [0.0 to 97.5] | 63.6 [30.8 to 89.1] | 33.3 [0.8 to 90.6] | 16.7 [0.4 to 64.1]

6. Secondary Outcome: CP-CML, AP-CML, BP-CML, and Ph+ALL Participants: Percentage of Participants With Major Molecular Response (MMR)
Description: MMR was defined as a ratio of reverse transcribed transcript of BCR-ABL to ABL <=0.1% on the International scale (equivalent to a 3-log reduction in transcript). Participants were non-responders in any of the following situations: BCR-ABL or ABL levels not detectable at baseline, no valid baseline or post-baseline assessment, and baseline assessment for e1a2 variant only.
Time Frame: Baseline up to 60 months
Population: Treated population included all participants who had received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ponatinib 30 mg: Phase 1 CP-CML | Ponatinib 30 mg: Phase 1 AP-CML | Ponatinib 30 mg: Phase 1 Ph+ ALL | Ponatinib 45 mg: Phase 1 CP-CML | Ponatinib 45 mg: Phase 1 AP-CML | Ponatinib 45 mg: Phase 1 BP-CML | Ponatinib 45 mg: Phase 1 Ph+ ALL | Ponatinib 15 mg: Phase 2 CP-CML | Ponatinib 15 mg: Phase 2 Ph+ ALL | Ponatinib 45 mg: Phase 2 CP-CML | Ponatinib 45 mg: Phase 2 BP-CML | Ponatinib 45 mg: Phase 2 PH+ ALL
Number analyzed (Participants) | 1 | 1 | 4 | 3 | 1 | 1 | 1 | 2 | 1 | 11 | 3 | 6
percentage of participants | 0 [0.0 to 97.5] | 0 [0.0 to 97.5] | 0 [0.0 to 60.2] | 100 [29.2 to 100] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5] | 50.0 [1.3 to 98.7] | 9 [0.0 to 97.5] | 27.3 [6.0 to 61.0] | 33.3 [0.8 to 90.6] | 0 [0.0 to 45.9]

7. Secondary Outcome: CP-CML, AP-CML, BP-CML, and Ph+ALL Participants: Median Time to Response (TTR)
Description: Time to response was defined as the interval from the first dose of study treatment until the criteria for response were first met, censored at the last assessment of response. Median time to response was estimated by Kaplan-Meier method.
Time Frame: From the first dose of study treatment until the criteria for response were first met (up to 60 months)
Population: Treated population included all participants who had received at least 1 dose of study drug.
Measure: Median (Full Range); unit: days
Arm/Group | Ponatinib 30 mg: Phase 1 CP-CML | Ponatinib 30 mg: Phase 1 AP-CML | Ponatinib 30 mg: Phase 1 Ph+ ALL | Ponatinib 45 mg: Phase 1 CP-CML | Ponatinib 45 mg: Phase 1 AP-CML | Ponatinib 45 mg: Phase 1 BP-CML | Ponatinib 45 mg: Phase 1 Ph+ ALL | Ponatinib 15 mg: Phase 2 CP-CML | Ponatinib 15 mg: Phase 2 Ph+ ALL | Ponatinib 45 mg: Phase 2 CP-CML | Ponatinib 45 mg: Phase 2 BP-CML | Ponatinib 45 mg: Phase 2 PH+ ALL
Number analyzed (Participants) | 1 | 1 | 4 | 3 | 1 | 1 | 1 | 2 | 2 | 11 | 3 | 6
days
  Cytogenic response | 85.0 [85 to 85] | NA [NA to NA] — Median and 95% CI were not estimable as excessive participants were censored. | NA [NA to NA] — Median and 95% CI were not estimable as excessive participants were censored. | 85 [85 to 169] | 113 [113 to 113] | 29 [29 to 29] | 28 [28 to 28] | 84 [84 to 84] | NA [NA to NA] — Median and 95% CI were not estimable as excessive participants were censored. | 167 [84 to 755] | 31 [31 to 31] | 29 [24 to 58]
  Hematologic response | NA [NA to NA] — Median and 95% CI were not estimable as excessive participants were censored. | 22 [22 to 22] | 14.5 [14 to 15] | NA [NA to NA] — Median and 95% CI were not estimable as excessive participants were censored. | 56 [56 to 56] | 15 [15 to 15] | NA [NA to NA] — Median and 95% CI were not estimable as excessive participants were censored. | NA [NA to NA] — Median and 95% CI were not estimable as excessive participants were censored. | NA [NA to NA] — Median and 95% CI were not estimable as excessive participants were censored. | NA [NA to NA] — Median and 95% CI were not estimable as excessive participants were censored. | 17 [17 to 17] | 15 [10 to 44]
  Molecular response | NA [NA to NA] — Median and 95% CI were not estimable as excessive participants were censored. | NA [NA to NA] — Median and 95% CI were not estimable as excessive participants were censored. | NA [NA to NA] — Median and 95% CI were not estimable as excessive participants were censored. | 85 [85 to 421] | NA [NA to NA] — Median and 95% CI were not estimable as excessive participants were censored. | NA [NA to NA] — Median and 95% CI were not estimable as excessive participants were censored. | NA [NA to NA] — Median and 95% CI were not estimable as excessive participants were censored. | 84 [84 to 84] | NA [NA to NA] — Median and 95% CI were not estimable as excessive participants were censored. | 253.0 [84 to 842] | 58 [58 to 58] | NA [NA to NA] — Median and 95% CI were not estimable as excessive participants were censored.

8. Secondary Outcome: CP-CML and Advanced Phase Participants: Median Duration of Response (DOR)
Description: DOR: interval between first assessment at which criteria for response was met, until criteria for progression was met, censored at last date at which criteria for response was met. DOR was estimated using the Kaplan-Meier method. Progression criteria for CP was: death, development of AP/BP, or loss of CHR (in absence of cytogenic response), or loss of MCyR, or increasing WBC in participant without CHR (doubling of WBCs to >20,000 on 2 occasions at least 4 weeks apart, after first week of therapy), as confirmed by development in complete blood cells (CBCs) at least 4 weeks apart; AP was: death, development of confirmed BP, loss of previous major/minor hematologic response over-2 week period, or no decrease from baseline levels in percentage blasts in peripheral blood/BM on all assessments over a 4-week period; and BP/Ph+ALL was: death/increasing blasts in peripheral blood or BM over a 4-week period. As planned, DOR is reported for all participants by entry mutation (T315I and Other).
Time Frame: From the first assessment at which criteria for response was met until the criteria for progression was first met (up to 60 months)
Population: Treated population by entry mutation. Here number analyzed "n" are the participants who were evaluable for this outcome measure for given categories.
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Ponatinib 30 mg: Phase 1 CP-CML Participants With T315I Mutations: Ponatinib 30 mg, tablet, orally, once daily in a 28-day treatment cycle for up to unacceptable drug reaction or disease progression (up to 60 months) in participants with CP-CML resistant or intolerant to dasatinib or nilotinib and who had (T)hreonine-315-(I)soleucine mutation (T315I) mutation of BCR-ABL in Dose-escalation Phase 1.
- Ponatinib 45 mg: Phase 1 CP-CML Participants With T315I Mutations: Ponatinib 45 mg, tablet, orally, once daily in a 28-day treatment cycle for up to unacceptable drug reaction or disease progression (up to 60 months) in participants with CP-CML resistant or intolerant to dasatinib or nilotinib and who had T315I mutation of BCR-ABL in Dose-escalation Phase 1.
- Ponatinib 15 mg: Phase 2 CP-CML Participants With T315I Mutations: Ponatinib 15 mg, tablet, orally, once daily for 7-days in a 28-day treatment cycle in participants with CP-CML resistant or intolerant to dasatinib or nilotinib and who had T315I mutation of BCR-ABL in Expansion Phase 2. Dose was increased to ponatinib 45 mg in the same participants at the discretion of Investigator and was administered as tablet, orally, once daily in a 28-day treatment Cycle for up to unacceptable drug reaction or disease progression (up to 60 months).
- Ponatinib 45 mg: Phase 2 CP-CML Participants With T315I Mutations: Ponatinib 45 mg, tablet, orally, once daily in a 28-day treatment cycle for up to unacceptable drug reaction or disease progression (up to 60 months) in participants with CP-CML resistant or intolerant to dasatinib or nilotinib and who had T315I mutation of BCR-ABL in Expansion Phase 2.
- Ponatinib 30 mg: Phase 1 CP-CML Participants With Other Mutations: Ponatinib 30 mg, tablet, orally, once daily in a 28-day treatment cycle for up to unacceptable drug reaction or disease progression (up to 60 months) in participants CP-CML resistant or intolerant to dasatinib or nilotinib and who had mutation other than T315I, no mutations, and no sequencing data in Dose-escalation Phase 1.
- Ponatinib 45 mg: Phase 1 CP-CML Participants With Other Mutations: Ponatinib 45 mg, tablet, orally, once daily in a 28-day treatment cycle for up to unacceptable drug reaction or disease progression (up to 60 months) in participants with CP-CML resistant or intolerant to dasatinib or nilotinib and who had mutation other than T315I, no mutations, and no sequencing data in Dose-escalation Phase 1.
- Ponatinib 15 mg: Phase 2 CP-CML Participants With Other Mutations: Ponatinib 15 mg, tablet, orally, once daily for 7-days in a 28-day treatment cycle in participants with CP-CML resistant or intolerant to dasatinib or nilotinib and who had mutation other than T315I, no mutations, and no sequencing data in Expansion Phase 2. Dose was increased to ponatinib 45 mg in the same participants at the discretion of Investigator and was administered as tablet, orally, once daily in a 28-day treatment cycle for up to unacceptable drug reaction or disease progression (up to 60 months).
- Ponatinib 45 mg: Phase 2 CP-CML Participants With Other Mutations: Ponatinib 45 mg, tablet, orally, once daily in a 28-day treatment cycle for up to unacceptable drug reaction or disease progression (up to 60 months) in participants with CP-CML resistant or intolerant to dasatinib or nilotinib and who had mutation other than T315I, no mutations, and no sequencing data in Expansion Phase 2.
- Ponatinib 30 mg: Phase 1 Advanced Phase Participants With T315I Mutations: Ponatinib 30 mg, tablet, orally, once daily in a 28-day treatment cycle for up to unacceptable drug reaction or disease progression (up to 60 months) in participants with AP-CML and BP-CML resistant or intolerant to dasatinib or nilotinib and Ph+ ALL participants and who had T315I mutation of BCR-ABL in Dose-escalation Phase 1.
- Ponatinib 45 mg: Phase 1 Advanced Phase Participants With T315I Mutations: Ponatinib 45 mg, tablet, orally, once daily in a 28-day treatment cycle for up to unacceptable drug reaction or disease progression (up to 60 months) in participants with AP-CML and BP-CML resistant or intolerant to dasatinib or nilotinib and Ph+ ALL participants and who had T315I mutation of BCR-ABL in Dose-escalation Phase 1.
- Ponatinib 15 mg: Phase 2 Advanced Phase Participants With T315I Mutations: Ponatinib 15 mg, tablet, orally, once daily in a 28-day treatment cycle for up to unacceptable drug reaction or disease progression (up to 60 months) in participants with AP-CML and BP-CML resistant or intolerant to dasatinib or nilotinib and Ph+ ALL participants and who had T315I mutation of BCR-ABL in Expansion Phase 2.
- Ponatinib 45 mg: Phase 2 Advanced Phase Participants With T315I Mutations: Ponatinib 45 mg, tablet, orally, once daily in a 28-day treatment cycle for up to unacceptable drug reaction or disease progression (up to 60 months) in participants with AP-CML and BP-CML resistant or intolerant to dasatinib or nilotinib and Ph+ ALL participants and who had T315I mutation of BCR-ABL in Expansion Phase 2.
- Ponatinib 30 mg: Phase 1 Advanced Phase Participants With Other Mutations: Ponatinib 30 mg, tablet, orally, once daily in a 28-day treatment cycle for up to unacceptable drug reaction or disease progression (up to 60 months) in participants with AP-CML and BP-CML resistant or intolerant to dasatinib or nilotinib and Ph+ ALL participants and who had mutation other than T315I, no mutations, and no sequencing data in Dose-escalation Phase 1.
- Ponatinib 45 mg: Phase 1 Advanced Phase Participants With Other Mutations: Ponatinib 45 mg, tablet, orally, once daily in a 28-day treatment cycle for up to unacceptable drug reaction or disease progression (up to 60 months) in participants with AP-CML and BP-CML resistant or intolerant to dasatinib or nilotinib and Ph+ ALL participants and who had mutation other than T315I, no mutations, and no sequencing data in Dose-escalation Phase 1.
- Ponatinib 15 mg: Phase 2 Advanced Phase Participants With Other Mutations: Ponatinib 15 mg, tablet, orally, once daily in a 28-day treatment cycle for up to unacceptable drug reaction or disease progression (up to 60 months) in participants with AP-CML and BP-CML resistant or intolerant to dasatinib or nilotinib and Ph+ ALL participants and who had mutation other than T315I, no mutations, and no sequencing data in Expansion Phase 2.
- Ponatinib 45 mg: Phase 2 Advanced Phase Participants With Other Mutations: Ponatinib 45 mg, tablet, orally, once daily in a 28-day treatment cycle for up to unacceptable drug reaction or disease progression (up to 60 months) in participants with AP-CML and BP-CML resistant or intolerant to dasatinib or nilotinib and Ph+ ALL participants and who had mutation other than T315I, no mutations, and no sequencing data in Expansion Phase 2.
Arm/Group | Ponatinib 30 mg: Phase 1 CP-CML Participants With T315I Mutations | Ponatinib 45 mg: Phase 1 CP-CML Participants With T315I Mutations | Ponatinib 15 mg: Phase 2 CP-CML Participants With T315I Mutations | Ponatinib 45 mg: Phase 2 CP-CML Participants With T315I Mutations | Ponatinib 30 mg: Phase 1 CP-CML Participants With Other Mutations | Ponatinib 45 mg: Phase 1 CP-CML Participants With Other Mutations | Ponatinib 15 mg: Phase 2 CP-CML Participants With Other Mutations | Ponatinib 45 mg: Phase 2 CP-CML Participants With Other Mutations | Ponatinib 30 mg: Phase 1 Advanced Phase Participants With T315I Mutations | Ponatinib 45 mg: Phase 1 Advanced Phase Participants With T315I Mutations | Ponatinib 15 mg: Phase 2 Advanced Phase Participants With T315I Mutations | Ponatinib 45 mg: Phase 2 Advanced Phase Participants With T315I Mutations | Ponatinib 30 mg: Phase 1 Advanced Phase Participants With Other Mutations | Ponatinib 45 mg: Phase 1 Advanced Phase Participants With Other Mutations | Ponatinib 15 mg: Phase 2 Advanced Phase Participants With Other Mutations | Ponatinib 45 mg: Phase 2 Advanced Phase Participants With Other Mutations
Number analyzed (Participants) | 1 | 0 | 0 | 1 | 0 | 3 | 2 | 9 | 2 | 2 | 0 | 4 | 1 | 1 | 0 | 2
days
  Cytogenic response: number analyzed (Participants) | 1 | 0 | 0 | 1 | 0 | 3 | 1 | 6 | 0 | 2 | 0 | 4 | 0 | 1 | 0 | 1
  Cytogenic response | 1513.0 [NA to NA] — 95% CI were not estimable as excessive participants were censored. |  |  | NA [NA to NA] — Median and 95% CI were not estimable as excessive participants were censored. |  | NA [NA to NA] — Median and 95% CI were not estimable as excessive participants were censored. | NA [NA to NA] — Median and 95% CI were not estimable as excessive participants were censored. | NA [NA to NA] — Median and 95% CI were not estimable as excessive participants were censored. |  | NA [NA to NA] — Median and 95% CI were not estimable as excessive participants were censored. |  | 31.0 [20.0 to NA] — 95% CI (upper limit) were not estimable as excessive participants were censored. |  | 169.0 [NA to NA] — 95% CI were not estimable as excessive participants were censored. |  | 205.0 [NA to NA] — 95% CI were not estimable as excessive participants were censored.
  Hematologic response: number analyzed (Participants) | 1 | 0 | 0 | 1 | 0 | 3 | 2 | 9 | 2 | 1 | 0 | 4 | 1 | 1 | 0 | 2
  Hematologic response | NA [NA to NA] — Median and 95% CI were not estimable as excessive participants were censored. |  |  | NA [NA to NA] — Median and 95% CI were not estimable as excessive participants were censored. |  | NA [1226.0 to NA] — Median and 95% CI (upper limit) were not estimable as excessive participants were censored. | NA [NA to NA] — Median and 95% CI were not estimable as excessive participants were censored. | NA [85.0 to NA] — Median and 95% CI (upper limit) were not estimable as excessive participants were censored. | 56.5 [38.0 to NA] — 95% CI (upper limit) were not estimable as excessive participants were censored. | NA [NA to NA] — Median and 95% CI were not estimable as excessive participants were censored. |  | 50.5 [33.0 to NA] — 95% CI (upper limit) were not estimable as excessive participants were censored. | NA [NA to NA] — Median and 95% CI were not estimable as excessive participants were censored. | 226.0 [NA to NA] — 95% CI were not estimable as excessive participants were censored. |  | 113.5 [110.0 to NA] — 95% CI (upper limit) were not estimable as excessive participants were censored.
  Molecular response: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Molecular response |  |  |  | NA [NA to NA] — Median and 95% CI were not estimable as excessive participants were censored. |  | NA [NA to NA] — Median and 95% CI were not estimable as excessive participants were censored. | NA [NA to NA] — Median and 95% CI were not estimable as excessive participants were censored. | NA [NA to NA] — Median and 95% CI were not estimable as excessive participants were censored. |  |  |  | 168.0 [NA to NA] — 95% CI were not estimable as excessive participants were censored. |  |  |  |

9. Secondary Outcome: CP-CML and Advanced Phase Participants: Median Progression-free Survival (PFS)
Description: PFS: interval from the first dose of study treatment until the criteria for progression or death were met, censored at the last response assessment. PFS was estimated using the Kaplan-Meier method. Progression criteria for CP was: death, development of AP/BP, or loss of CHR (in absence of cytogenic response), or loss of MCyR, or increasing WBC in participant without CHR (doubling of WBCs to >20,000 on 2 occasions at least 4 weeks apart, after first week of therapy), as confirmed by development in CBCs at least 4 weeks apart; AP was: death, development of confirmed BP, loss of previous major/minor hematologic response over-2 week period, or no decrease from baseline levels in percentage blasts in peripheral blood/BM on all assessments over a 4-week period; BP/Ph+ALL was: death or increasing blasts in peripheral blood or BM over a 4-week period. As planned, PFS is reported for all participants by entry mutation (T315I and Other).
Time Frame: From the first assessment at which criteria for response was met until the criteria for progression or death was met (up to 60 months)
Population: Treated population by entry mutation. Here overall number analyzed "N" are the participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Ponatinib 30 mg: Phase 1 CP-CML Participants With T315I Mutations: Ponatinib 30 mg, tablet, orally, once daily in a 28-day treatment cycle for up to unacceptable drug reaction or disease progression (up to 60 months) in participants with CP-CML resistant or intolerant to dasatinib or nilotinib and who had T315I mutation of BCR-ABL in Dose-escalation Phase 1.
- Phase 2: Ponatinib 45 mg, Advanced Phase Participants With Other Mutations: Ponatinib 45 mg, tablet, orally, once daily in a 28-day treatment Cycle for up to unacceptable drug reaction or disease progression (up to 60 months) in participants with AP-CML and BP-CML resistant or intolerant to dasatinib or nilotinib and Ph+ ALL participants and who had mutation other than T315I, no mutations, and no sequencing data in Expansion Phase 2.
Arm/Group | Ponatinib 30 mg: Phase 1 CP-CML Participants With T315I Mutations | Ponatinib 45 mg: Phase 1 CP-CML Participants With T315I Mutations | Ponatinib 15 mg: Phase 2 CP-CML Participants With T315I Mutations | Ponatinib 45 mg: Phase 2 CP-CML Participants With T315I Mutations | Ponatinib 30 mg: Phase 1 CP-CML Participants With Other Mutations | Ponatinib 45 mg: Phase 1 CP-CML Participants With Other Mutations | Ponatinib 15 mg: Phase 2 CP-CML Participants With Other Mutations | Ponatinib 45 mg: Phase 2 CP-CML Participants With Other Mutations | Ponatinib 30 mg: Phase 1 Advanced Phase Participants With T315I Mutations | Ponatinib 45 mg: Phase 1 Advanced Phase Participants With T315I Mutations | Ponatinib 15 mg: Phase 2 Advanced Phase Participants With T315I Mutations | Ponatinib 45 mg: Phase 2 Advanced Phase Participants With T315I Mutations | Ponatinib 30 mg: Phase 1 Advanced Phase Participants With Other Mutations | Ponatinib 45 mg: Phase 1 Advanced Phase Participants With Other Mutations | Ponatinib 15 mg: Phase 2 Advanced Phase Participants With Other Mutations | Phase 2: Ponatinib 45 mg, Advanced Phase Participants With Other Mutations
Number analyzed (Participants) | 1 | 0 | 0 | 2 | 0 | 3 | 2 | 9 | 3 | 2 | 1 | 5 | 2 | 1 | 0 | 4
days | 1597.0 [NA to NA] — 95% CI were not estimable as excessive participants were censored. |  |  | NA [85.0 to NA] — Median and 95% CI (upper limit) were not estimable as excessive participants were censored. |  | NA [NA to NA] — Median and 95% CI were not estimable as excessive participants were censored. | NA [NA to NA] — Median and 95% CI were not estimable as excessive participants were censored. | NA [113.0 to NA] — Median and 95% CI (upper limit) were not estimable as excessive participants were censored. | 51.0 [29.0 to NA] — 95% CI (upper limit) were not estimable as excessive participants were censored. | 320.0 [113.0 to NA] — 95% CI (upper limit) were not estimable as excessive participants were censored. | 33.0 [NA to NA] — 95% CI were not estimable as excessive participants were censored. | 100.0 [10.0 to NA] — 95% CI (upper limit) were not estimable as excessive participants were censored. | 56.5 [10.0 to NA] — 95% CI (upper limit) were not estimable as excessive participants were censored. | 281.0 [NA to NA] — 95% CI were not estimable as excessive participants were censored. |  | 127.5 [85.0 to NA] — 95% CI (upper limit) were not estimable as excessive participants were censored.

10. Secondary Outcome: CP-CML and Advanced Phase Participants: Overall Survival (OS)
Description: OS was defined as the interval from the first dose of study treatment until death, censored at the last date at which participant was known to be alive. Overall survival was estimated using the Kaplan-Meier method. As planned, OS is reported for all participants by entry mutation (T315I and Other).
Time Frame: From the first dose of study treatment until death (up to 60 months)
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Ponatinib 30 mg: Phase 1 Ponatinib 30 mg: Phase 1 Advanced Phase Participants With T315I Mutations: Ponatinib 30 mg, tablet, orally, once daily in a 28-day treatment cycle for up to unacceptable drug reaction or disease progression (up to 60 months) in participants with AP-CML and BP-CML resistant or intolerant to dasatinib or nilotinib and Ph+ ALL participants and who had T315I mutation of BCR-ABL in Dose-escalation Phase 1.
Arm/Group | Ponatinib 30 mg: Phase 1 CP-CML Participants With T315I Mutations | Ponatinib 45 mg: Phase 1 CP-CML Participants With T315I Mutations | Ponatinib 15 mg: Phase 2 CP-CML Participants With T315I Mutations | Ponatinib 45 mg: Phase 2 CP-CML Participants With T315I Mutations | Ponatinib 30 mg: Phase 1 CP-CML Participants With Other Mutations | Ponatinib 45 mg: Phase 1 CP-CML Participants With Other Mutations | Ponatinib 15 mg: Phase 2 CP-CML Participants With Other Mutations | Ponatinib 45 mg: Phase 2 CP-CML Participants With Other Mutations | Ponatinib 30 mg: Phase 1 Ponatinib 30 mg: Phase 1 Advanced Phase Participants With T315I Mutations | Ponatinib 45 mg: Phase 1 Advanced Phase Participants With T315I Mutations | Ponatinib 15 mg: Phase 2 Advanced Phase Participants With T315I Mutations | Ponatinib 45 mg: Phase 2 Advanced Phase Participants With T315I Mutations | Ponatinib 30 mg: Phase 1 Advanced Phase Participants With Other Mutations | Ponatinib 45 mg: Phase 1 Advanced Phase Participants With Other Mutations | Ponatinib 15 mg: Phase 2 Advanced Phase Participants With Other Mutations | Ponatinib 45 mg: Phase 2 Advanced Phase Participants With Other Mutations
Number analyzed (Participants) | 1 | 0 | 0 | 2 | 0 | 3 | 2 | 9 | 3 | 2 | 1 | 5 | 2 | 1 | 0 | 4
days | NA [NA to NA] — Median and 95% CI were not estimable as excessive participants were censored. |  |  | NA [NA to NA] — Median and 95% CI were not estimable as excessive participants were censored. |  | NA [NA to NA] — Median and 95% CI were not estimable as excessive participants were censored. | NA [NA to NA] — Median and 95% CI were not estimable as excessive participants were censored. | NA [1305.0 to NA] — Median and 95% CI (upper limit) were not estimable as excessive participants were censored. | 201.0 [194.0 to NA] — 95% CI (upper limit) were not estimable as excessive participants were censored. | NA [527.0 to NA] — Median and 95% CI (upper limit) were not estimable as excessive participants were censored. | 109.0 [NA to NA] — 95% CI were not estimable as excessive participants were censored. | 264.0 [169.0 to NA] — 95% CI (upper limit) were not estimable as excessive participants were censored. | 131.0 [10.0 to NA] — 95% CI (upper limit) were not estimable as excessive participants were censored. | 382.0 [NA to NA] — 95% CI were not estimable as excessive participants were censored. |  | 550.5 [281.0 to NA] — 95% CI (upper limit) were not estimable as excessive participants were censored.

11. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for Ponatinib
Time Frame: Cycle 1 Day 1 pre-dose and at multiple time points (up to 24 hours) post-dose (Cycle length= 28 days)
Population: Treated population include all participants who had received at least 1 dose of study drug and for whom PK samples were collected. As planned, PK samples were analyzed per dose level.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Groups:
- Ponatinib 15 mg: Ponatinib 15 mg, tablet, orally, once daily for 7-days in a 28-day treatment Cycle 1 before 15 mg was dose-escalated to recommended phase 2 dose (RP2D) in participants with CP-CML, BP-CML, or AP-CML who were resistant or intolerant to dasatinib or nilotinib, or with Ph+ALL who were resistant or intolerant to prior TKIs.
- Ponatinib 30 mg: Ponatinib 30 mg, tablet, orally, once daily in a 28-day treatment Cycle 1 in participants with CP-CML, BP-CML, or AP-CML who were resistant or intolerant to dasatinib or nilotinib, or with Ph+ALL who were resistant or intolerant to prior TKIs.
- Ponatinib 45 mg: Ponatinib 45 mg, tablet, orally, once daily in a 28-day treatment Cycle 1 in participants with CP-CML, BP-CML, or AP-CML who were resistant or intolerant to dasatinib or nilotinib, or with Ph+ALL who were resistant or intolerant to prior TKIs.
Arm/Group | Ponatinib 15 mg | Ponatinib 30 mg | Ponatinib 45 mg
Number analyzed (Participants) | 3 | 6 | 6
nanogram per milliliter (ng/mL) | 23.67 (7.136) | 31.55 (9.072) | 89.13 (24.63)

12. Secondary Outcome: Tmax: Time to Reach the Cmax for Ponatinib
Time Frame: Cycle 1 Day 1 pre-dose and at multiple time points (up to 24 hours) post-dose (Cycle length= 28 days)
Population: as for outcome 11
Measure: Median (Full Range); unit: hour
Groups:
- Ponatinib 15 mg: Ponatinib 15 mg, tablet, orally, once daily for 7-days in a 28-day treatment Cycle 1 before 15 mg was dose-escalated to RP2D in participants with CP-CML, BP-CML, or AP-CML who were resistant or intolerant to dasatinib or nilotinib, or with Ph+ALL who were resistant or intolerant to prior TKIs.
Arm/Group | Ponatinib 15 mg | Ponatinib 30 mg | Ponatinib 45 mg
Number analyzed (Participants) | 3 | 6 | 6
hour | 4.00 [4.0 to 6.2] | 6.75 [3.9 to 8.1] | 5.00 [4.0 to 6.0]

13. Secondary Outcome: AUC(0-24): Area Under the Plasma Concentration-time Curve From Time 0 to 24 Hours Post-dose for Ponatinib
Time Frame: Cycle 1 Day 1 pre-dose and at multiple time points (up to 24 hours) post-dose (Cycle length= 28 days)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Ponatinib 15 mg | Ponatinib 30 mg | Ponatinib 45 mg
Number analyzed (Participants) | 3 | 6 | 6
hour*nanogram per milliliter (h*ng/mL) | 336.00 (129.55) | 495.98 (154.09) | 1385.5 (456.20)

14. Secondary Outcome: T1/2: Terminal Phase Elimination Half-life for Ponatinib
Time Frame: Cycle 1 Day 1 pre-dose and at multiple time points (up to 24 hours) post-dose (Cycle length= 28 days)
Population: as for outcome 11
Measure: Median (Full Range); unit: hours
Arm/Group | Ponatinib 15 mg | Ponatinib 30 mg | Ponatinib 45 mg
Number analyzed (Participants) | 3 | 6 | 6
hours | NA [NA to NA] — Data could not be calculated for t1/2 due to lack of PK time points beyond 24 hours post-dose. | NA [NA to NA] — Data could not be calculated for t1/2 due to lack of PK time points beyond 24 hours post-dose. | NA [NA to NA] — Data could not be calculated for t1/2 due to lack of PK time points beyond 24 hours post-dose.

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) are AEs that started after the first dose of study drug up to 5 years and 11 months
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Ponatinib 30 mg: Phase 1 CP-CML | Ponatinib 30 mg: Phase 1 AP-CML | Ponatinib 30 mg: Phase 1 Ph+ ALL | Ponatinib 45 mg: Phase 1 CP-CML | Ponatinib 45 mg: Phase 1 AP-CML | Ponatinib 45 mg: Phase 1 BP-CML | Ponatinib 45 mg: Phase 1 Ph+ ALL | Ponatinib 15 mg: Phase 2 CP-CML | Ponatinib 15 mg: Phase 2 Ph+ ALL | Ponatinib 45 mg: Phase 2 CP-CML | Ponatinib 45 mg: Phase 2 BP-CML | Ponatinib 45 mg: Phase 2 PH+ ALL
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 4/4 | 0/3 | 1/1 | 0/1 | 1/1 | 0/2 | 1/1 | 1/11 | 3/3 | 6/6
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/1 | 2/4 | 2/3 | 1/1 | 0/1 | 0/1 | 1/2 | 1/1 | 6/11 | 2/3 | 1/6
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 3/4 | 3/3 | 1/1 | 1/1 | 1/1 | 2/2 | 1/1 | 11/11 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ponatinib 30 mg: Phase 1 CP-CML (N=1) | Ponatinib 30 mg: Phase 1 AP-CML (N=1) | Ponatinib 30 mg: Phase 1 Ph+ ALL (N=4) | Ponatinib 45 mg: Phase 1 CP-CML (N=3) | Ponatinib 45 mg: Phase 1 AP-CML (N=1) | Ponatinib 45 mg: Phase 1 BP-CML (N=1) | Ponatinib 45 mg: Phase 1 Ph+ ALL (N=1) | Ponatinib 15 mg: Phase 2 CP-CML (N=2) | Ponatinib 15 mg: Phase 2 Ph+ ALL (N=1) | Ponatinib 45 mg: Phase 2 CP-CML (N=11) | Ponatinib 45 mg: Phase 2 BP-CML (N=3) | Ponatinib 45 mg: Phase 2 PH+ ALL (N=6)
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enteritis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia legionella (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetic nephropathy (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Brain stem infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Genital haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retinal vein occlusion (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mechanical ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ponatinib 30 mg: Phase 1 CP-CML (N=1) | Ponatinib 30 mg: Phase 1 AP-CML (N=1) | Ponatinib 30 mg: Phase 1 Ph+ ALL (N=4) | Ponatinib 45 mg: Phase 1 CP-CML (N=3) | Ponatinib 45 mg: Phase 1 AP-CML (N=1) | Ponatinib 45 mg: Phase 1 BP-CML (N=1) | Ponatinib 45 mg: Phase 1 Ph+ ALL (N=1) | Ponatinib 15 mg: Phase 2 CP-CML (N=2) | Ponatinib 15 mg: Phase 2 Ph+ ALL (N=1) | Ponatinib 45 mg: Phase 2 CP-CML (N=11) | Ponatinib 45 mg: Phase 2 BP-CML (N=3) | Ponatinib 45 mg: Phase 2 PH+ ALL (N=6)
Platelet count decreased (Investigations) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 7 | 0 | 2
Lipase increased (Investigations) | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 3 | 1 | 3
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 3
Alanine aminotransferase increased (Investigations) | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 4 | 2 | 2
Weight decreased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Amylase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Weight increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Blood uric acid increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood creatine phosphokinase decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood phosphorus increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Brain natriuretic peptide increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram t wave inversion (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypotension (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Protein C decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urine output decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 4
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 2 | 0 | 2 | 2 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Asteatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 2 | 1 | 6 | 3 | 5
Oedema peripheral (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 3
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hyperthermia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 2 | 0 | 1 | 1 | 0 | 0 | 2 | 1 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 3 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Angular cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chronic gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 (0) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 (0) | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth loss (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Platelet count decreased (Blood and lymphatic system disorders) | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 3 | 2 | 1
Neutrophil count decreased (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 2
White blood cell count decreased (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctivitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Impetigo (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ophthalmic herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 (0) | 0 | 1 | 0 | 0
Perirectal abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyoderma (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinea infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Blood cholesterol increased (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypouricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Steroid diabetes (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 6 | 1 | 3
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Peripheral coldness (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebral artery occlusion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dementia alzheimers type (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hemiplegia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Parkinsons disease (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Trigeminal neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertensive nephropathy (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urethral pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Cystitis radiation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural inflammation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth avulsion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
CONJUNCTIVITIS allergic (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Corneal disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Macular degeneration (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uveitis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 1
Anxiety disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac aneurysm (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac discomfort (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood bilirubin increased (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Menstrual disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2013-11-21): https://cdn.clinicaltrials.gov/large-docs/33/NCT01667133/Prot_000.pdf
  • Statistical Analysis Plan (2015-03-04): https://cdn.clinicaltrials.gov/large-docs/33/NCT01667133/SAP_001.pdf